CLINICAL TRIAL: NCT06953908
Title: The Copenhagen Gender Identity Cohort
Acronym: KIK
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christina Esmann Fonvig, Research associate, Rigshospitalet, Denmark
Other Study IDs: 001
Record Dates: First submitted 2025-04-03; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Gender Identity; Gender Dysphoria, Adult; Gender Incongruence
Keywords: Gender Identity; Gender Incongruence
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults seeking help regarding gender incongruence: All patients referred to The Center of Gender Identity in Copenhagen (CGI), 18 years or older, seeking medical og surgical treatment for gender incongruence.

SUMMARY:
The goal of this observational study is to systematically collect data on adults seeking medical and surgical treatments for gender incongruence. This prospective, longitudinal cohort aims to generate insights into the safety, effectiveness, and overall satisfaction with current treatments. Additionally, the study seeks to identify areas for improvement and support healthcare professionals in making informed decisions. Most importantly, it aims to enhance the quality of life for transgender and gender-diverse individuals by ensuring that the care they receive aligns with their needs and goals.

Participants will include patients seeking treatment at the Copenhagen Center for Gender Identity, Denmark. Data collection will be both clinician- and patient-reported. Participants will be asked to complete online surveys at baseline, after the assessment process, and annually if they initiate hormone therapy. The study will systematically gather information on gender identity and transition experiences, sociodemographics, self-medication, health status, self-reported quality of life, and treatment preferences. Additionally, detailed records of treatment courses and specific interventions will be collected from all involved healthcare providers across specialties.

The study will evaluate the effects of different treatment options, both in the short and long term. It will explore how quality of life is associated with gender identity, transition, sociodemographics, lifestyle, and health, as well as assess the medical impact of various treatments, including counseling, hormone therapy, and surgery. Furthermore, the study will investigate the prevalence of side effects and complications related to treatment, as well as factors influencing treatment discontinuation, including cases of detransition.

Finally, the project will focus on quality indicators such as waiting times and patient satisfaction, contributing to the ongoing development of high-quality, patient-centered care for transgender and gender-diverse individuals.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to The Center for Gender Identity in Copenhagen

Exclusion Criteria:

* Inability to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants must be deemed eligible for assessment at The Center for Gender Identity in Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2032-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of quality of life | Baseline and latest yearly assessment.
  The study uses the WHOQOL-BREF to assesses quality of life (QOL). The repeated assessment provides a snapshot of quality of life, allowing for the exploration of associations with other factors. The WHOQOL-BREF is scored from 0-100, with higher values indicating increased quality of life.
  Change from baseline in the four domains (Physical Helath, Psychological, Relationships, Environment) to the latest recorded yearly assessment recorded within the study period (10 years from 2022-2032)

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Gender Identity, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data (IPD) is in conflict with Danish GDPR regulations, as it involves the transfer of personal and potentially sensitive information, which is restricted under Danish data protection laws to safeguard individuals' privacy and ensure compliance with strict legal and ethical requirements.